CLINICAL TRIAL: NCT03151096
Title: Pilot Evaluation of the Effect of Riboflavin Supplementation on Blood Pressure and Possible Effect Modification by the MTHFR C677T Genotype
Acronym: RiboBP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The target population with available genotype traveled outside study area and study duration of 19 weeks was long for some participants.
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: University of Ulster (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCC1518
Record Dates: First submitted 2017-04-18; First posted 2017-05-12 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: High Blood Pressure; MTHFR C677T Genotype
MeSH Terms: conditions — Hypertension | interventions — Riboflavin

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Field nurse measuring blood pressure, laboratory and data entry staff will be blinded as to the genotype of the study participants and to the identity of the treatment arm to which a participant is assigned from the time of randomization to the time of unblinding. The placebos are designed to be indistinguishable from the active drugs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment arm (Experimental): 5mg Riboflavin pills
  Interventions: Dietary Supplement: Riboflavin
- Placebo arm (Placebo Comparator): Placebo pills
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Riboflavin — one pill of Riboflavin will be taken orally with water
  Arms: treatment arm
Dietary Supplement: Placebo — one pill of placebo will be taken orally with water
  Arms: Placebo arm

SUMMARY:
Hypertension, which results from a combination of multiple lifestyle and genetic factors, is a global public health problem affecting 1 billion people worldwide. The identification of cheap treatment interventions without adverse side effects would be hugely advantageous particularly in low-income settings with high prevalence of hypertension such as sub-Saharan Africa where up to 46% of adults are affected.

Emerging evidence links a functional polymorphism in the MTHFR gene (rs1801133 C677T), encoding the folate-metabolising enzyme methylenetetrahydrofolate reductase to high blood pressure in adults. Variation at rs1801133 is relatively common and has 3 genotypes; homozygous "normal" CC, heterozygous CT and homozygous "variant" TT genotypes. Of these genotypes, the homozygous "variant" TT is more strongly associated with a higher BP. The precise mechanism by which MTHFR is associated with BP remains unclear. It has been recently shown in 3 separate randomized controlled trials that BP is highly responsive to riboflavin and that this response is differential by MTHFR rs1801133 genotype. In all these clinical trials, significant reduction in both systolic and diastolic blood pressure was observed in the homozygous variant TT genotype and an intermediate effect seen in those with the heterozygous CT genotype. The aim of this study is to evaluate the effect of riboflavin supplementation on blood pressure in a riboflavin-deplete population as well as comparing plasma riboflavin status before and after supplementation. This will be achieved by conducting a randomized single-blind placebo controlled trial over a period of 16 weeks.

The Investigators will use the Keneba biobank to invite about 100 adults with the CT genotype and a similar number of age-, sex and village-matched CC homozygotes. Participants within each of the groups will be randomized to receive either riboflavin (5mg/d) or a matching placebo which would be supplied on a weekly basis. Blood sample, blood pressure measurement, socio-demographic data and their anthropometric measurements (height, weight, waist and hip circumference and body composition by BIA) will be taken during the initial visit. An additional blood sample will be taken at the end of the study whilst additional BP measurements will be taken respectively at 8 weeks and at the end of the intervention. The possibility that riboflavin deficiency represents a new, easily-correctible causal factor in hypertension in sub-Saharan Africa would require further large-scale interventions if this pilot study yields encouraging results.

DETAILED DESCRIPTION:
This is a recall-by-genotype randomized single-blind placebo-controlled micronutrient supplementation trial. The Keneba biobank will be used to identify all potential participants i.e. individuals genotyped for MTHFR C677T for this pilot study.

The Investigators will invite all 163 adults with the CT genotype in the Keneba biobank and a similar number of age- sex- and village-matched CC homozygotes to participate in the study. Field assistants will visit the homes of potentially eligible participants, to provide full information about the purpose and methods of the study, potential risks and benefits, and participants' rights. Participants will then provide written informed consent. The field assistant will ensure that the conversation and consent process occurs in a private area or room, to maintain privacy and confidentiality. After exclusions and non-consenters the investigators anticipate at least 102 subjects per group. Using standard deviation estimates from our own and published literature (14mmHg for SBP and 10mmHg for DBP) the investigators will have 95% confidence (at p<0.05) of detecting differences of 3.88mmHg for SBP and 2.76mmHg for DBP.

Participants within each of the groups will be randomized to riboflavin or placebo in a 1:1 ratio according to a computer generated randomization scheme. This will be done by randomly assigning study numbers within the CT carriers to a treatment group and enrolling participants sequentially from lowest to highest study identification number. The subjects will be randomized upon dispensing the study drug associated with the subject pair's study identification number. Field, clinical, laboratory and data entry staff will be blinded to the genotype of the study participants and to the identity of the treatment arm to which a participant is assigned from the time of randomization to the time of unblinding. The placebos are designed to be indistinguishable from the active drugs. Double-blinding is not possible because subjects randomized to the riboflavin will have yellow urine (a harmless outcome that will be explained to them).

Eligible participants will then be invited for a visit to the MRC Keneba field station. At the initial visit, socio-demographic data and anthropometric measurements (height, weight, waist and hip circumference and body composition by BIA) will be taken. Thereafter, BP will be measured with an automated device in triplicate using a standard protocol by the same investigator who will be blinded to genotype and treatment group. The investigators will also collect 10ml sample of blood for laboratory assessment of vitamin B status. During the intervention phase of the trial, the investigators will supplement participants with 5mg/day of riboflavin or a matching placebo for 16 weeks. The pills will be supplied on a weekly basis with instructions to return any unused pills. Another BP measurement following similar protocol as before will be taken at 8 weeks as well as at 16 weeks after the start of the intervention. Finally, a 10ml blood sample will be collected at 16 weeks. Blood samples will be analysed for riboflavin, homocysteine, red cell folate, cobalamin and pyridoxine. Participants who were randomized to receive placebo will be offered riboflavin supplementation at the end of the study.

The investigators will use multilevel modeling test for a main effect of intervention on delta BP from baseline to 16wk (and repeated at 8wk) adjusted for sex and age. Chi-squared test will be used to test for changes in frequency of raised BP (>140/90). Then the investigators will test for effect modification according to MTHFR variant.

ELIGIBILITY:
Inclusion Criteria:

Healthy, aged between 18-70 years

* Has provided appropriate ethical consent for involvement in studies relating to genetics.
* Has available genotype data in the Keneba biobank needed for the current study
* Available for the duration of the intervention period

Exclusion Criteria:

Taking vitamin B/multivitamin supplements

* Ongoing pregnancy as confirmed by participant
* History of digestive, hepatic, renal or hematological disorders, dementia
* Epilepsy or taking anti-epileptic medications
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2019-04-22 (Actual); Study Completion 2019-04-22 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 16 weeks
  The aim of this study is to investigate whether supplementing 5mg of riboflavin can decrease blood pressure more effectively compared with placebo
Erythrocyte Glutathione Reductase Activation Coefficient (indicator of riboflavin status) | 16 weeks
  We will compare EGRAC in those who were randomised to riboflavin supplementation versus placebo

SECONDARY OUTCOMES:
Blood pressure | 16 weeks
  We would like to investigate if there is any effect modification in CC vs CT variants of rs1801133 in the MTHFR gene in response to riboflavin supplementation vs placebo
Blood pressure and plasma riboflavin status | 16 weeks
  We aim to describe the cross-sectional associations at baseline between blood pressure (continuous variable and proportion >140/90mm) and riboflavin status (assessed by the Erythrocyte Glutathione Reductase Activation Coefficient) and MTHFR variants

CONTACTS AND LOCATIONS:
Locations (1):
- MRC Clinic Keneba, Keneba, West Kiang, The Gambia

IPD SHARING:
Plan to Share IPD: No